CLINICAL TRIAL: NCT00902915
Title: Lenalidomide and Dexamethasone for Treatment of Patients With Acute Myeloma (Light Chain)-Induced Renal Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Austrian Forum Against Cancer (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LD
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Multiple Myeloma Light Chain Induced Renal Insufficiency
Keywords: multiple myeloma renal insufficiency
MeSH Terms: interventions — Lenalidomide; Dexamethasone

ARMS (1):
- Lenalidomide - Dexamethasone (Experimental)
  Interventions: Drug: lenalidomide plus dexamethasone

INTERVENTIONS:
Drug: lenalidomide plus dexamethasone — peroral application; lenalidomide dosage according to severity grade of renal failure.

SUMMARY:
The purpose of this study is to determine efficacy of lenalidomide and dexamethasone in the treatment of patients with acute Myeloma (light chain)-induced renal failure.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Age at least 18 years at the time of signing the informed consent form.
* MM (all stages) with acute light chain induced renal impairment
* Patients with previously unknown MM and acute light chain induced renal failure (GFR<50ml/min and serum creatinine minimum 2.0 mg/dL) and with further workup revealing light chain induced renal injury with MM as underlying cause.
* Patients with previously established MM and normal renal function (GFR ≥60ml/min and serum creatinine ≤1.2mg/dl) with progressive disease and acute (within 6 weeks) light chain induced renal failure (GFR<50ml/min and creatinine ≥ 2.0 mg/dL).
* Disease progression will be documented by one or more of the following criteria:

  * Increase in serum paraprotein by >25%, or increase of 50% of 24 hour urine paraprotein excretion
  * Hypercalcemia
  * Progression of bone lesions
  * Decrease in Hb>2g/dl within 4 weeks (not induced by cytotoxic drugs)
  * Increase in bone marrow plasma cell infiltration by > 25%
* All previous medical anti-myeloma therapy (excluding corticosteroids) must have been discontinued at least 3 weeks prior to treatment in this study.
* Able to adhere to the study visit schedule and other protocol requirements.
* Measurable serum or urine paraprotein
* Laboratory test results within these ranges:

  * Glomerular filtration rate < 50ml/min
  * Serum creatinine ≥ 2.0mg/dL
  * Absolute leukocyte count ≥ 1.5 x 10G/L
  * Platelet count minimum 75 x 10G/L if bone marrow plasma cell infiltration (BMPC) is ≥50% or minimum 30 x 10G/L if BMPC infiltration is <50%.
  * Total bilirubin minimum 1.5 mg/dL
  * AST (SGOT) and ALT (SGPT) not more than 2,5 x ULN
* Females of childbearing potential (FCBP) must:

  * Understand that the study medication could have an expected teratogenic risk
  * Agree to use, and be able to comply with, effective contraception without interruption, 4 weeks before starting study drug, throughout study drug therapy (including dose interruptions) and for 4 weeks after the end of study drug therapy, even if she has amenorrhea. This applies unless the subject commits to absolute and continued abstinence confirmed on a monthly basis. The following are effective methods of contraception: Implant, Levonorgestrel-releasing intrauterine system (IUS, Medroxyprogesterone acetate depot), Tubal sterilization, Sexual intercourse with a vasectomised male partner only; vasectomy must be confirmed by two negative semen analyses Ovulation inhibitory progesterone-only pills (i.e., desogestrel)
  * Agree to have a medically supervised pregnancy test with a minimum sensitivity of 25 mIU/ml not more than 3 days before the start of study medication once the subject has been on effective contraception for at least 4 weeks. This requirement also applies to women of childbearing potential who practice complete and continued abstinence.
  * Agree to have a medically supervised pregnancy test every 4 weeks including 4 weeks after the end of study treatment, except in the case of confirmed tubal sterilization. These tests should be performed not more than 3 days before the start of next treatment. This requirement also applies to women of childbearing potential who practice complete and continued abstinence.
* Male subjects must:

  * Agree to use condoms throughout study drug therapy, during any dose interruption and for 28 days after cessation of study therapy if their partner is of childbearing potential and has no contraception.
  * Agree not to donate semen during study drug therapy and for 28 days after end of study drug therapy.
* All subjects must agree not to share study medication with another person and to return all unused study drug to the investigator
* Disease free of prior malignancies for minimum of 3 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast
* Agree to take low molecular weight heparin as prophylactic anticoagulation.

Exclusion Criteria:

* Acute renal failure due to other causes than light-chain induced nephropathy such as NSAIRS, antibiotics, or other nephrotoxic drugs, or others.
* Acute renal failure due to hypercalcemia only, without excretion of nephrotoxic light chains.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Any prior use of lenalidomide
* Any anti-myeloma therapy within 3 weeks before day 1 of first cycle, with the exception of dexamethasone 40mg (maximum dose 160mg) or corticosteroid equivalent.
* Any other experimental drug or therapy within 3 weeks of baseline
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Known positive for HIV or infectious hepatitis, type A, B or C or evidence of any severe active or chronic infection.
* Clinical significant heart disease (NYHA status>2)
* Pregnant or breast feeding females
* Anamnesis of thromboembolic complications, such as stroke, myocardial infarction and pulmonary embolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
To determine the response rate (CR, VGPR, PR, MR, SD, and PD) To determine the renal response rate To determine the relation between category of myeloma response and improvement in GFR To determine the proportion of patients spared hemodialysis

SECONDARY OUTCOMES:
Progression Free Survival, Event Free Survival, Overall Survival; Toxicity, evaluated according to the NCCN toxicity scale (type, frequency, severity, and relationship of adverse events to study treatment).

CONTACTS AND LOCATIONS:
Locations (5):
- Austria (3):
  - LKH Salzburg, 3rd Med. Dept., Salzburg
  - Austrian Forum Against Cancer; 1st Med. Dept., Center for Hematology and Oncology, Wilhelminenspital, Montleartstrasse 37, Vienna
  - Clinic Wels-Grieskirchen, 4th Internal Dept., Wels
- Czechia (2):
  - Faculty Hospital Brno and Faculty of Medicine MU, Brno
  - Charles University Prague, Prague